CLINICAL TRIAL: NCT03852290
Title: Association of the C677T and A1298C MTHFR Polymorphisms With Chemotherapy Effectiveness Among Patients With Metastatic Colorectal Cancer
Brief Title: C677T and A1298C MTHFR Polymorphisms and Fluoropyrimidine Effectiveness in Metastatic Colon Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Universidad de Costa Rica (Other)
Collaborators: Universitat Autonoma de Barcelona (Other)
Responsible Party: Principal Investigator, Allan Ramos-Esquivel, Principal Investigator, Universidad de Costa Rica
Other Study IDs: R017-SABI-00126
Record Dates: First submitted 2019-02-19; First posted 2019-02-25 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Colon Cancer; MTHFR Gene Mutation; Chemotherapeutic Toxicity; Chemotherapy Effect
Keywords: Colon cancer; Fluoropyrimidine
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA extracted from blood samples and tumor tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fluoropyrimidines are the backbone of chemotherapy regimes used to treat metastatic colorectal cancer (CRC). These drugs act in different pathways of folate metabolism altering DNA synthesis mainly by inhibition of the tymidylate synthase. For this reaction the 5,10-methylenetetrahydrofolate acts as cofactor. It has been demonstrated that A1298C and C677T polymorphisms in the methylenetetrahydrofolate reductase (MTHFR) gene result in reduced enzyme activity that leads to reduced availability of this important cofactor. Hence, we hypothesized that the presence of these polymorphisms are related to the efficacy and toxicity of fluoropyrimidines in patients with CRC.

DETAILED DESCRIPTION:
Patients with metastatic colorectal cancer are invited to join this study at the start of treatment with any fluoropyrimidine used alone or in combination with oxaliplatin and/or irinotecan +/- bevacizumab, panitumumab or cetuximab. DNA extraction will be done from blood and tissue samples to determine the C677T (rs1801133) and 1298 A>C (rs18011131) polymorphisms of the MTHFR gene.

The patient will be followed at least for one year during treatment to determine any toxicity related to the therapy and to determine the overall survival, progression-free survival and response rate. Patients will be categorized into different categories according to the genetic status of each polymorphism.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic colorectal cancer receiving first line therapy with any fluoropyrimidine (capecitabine or 5-Fluorouracil) alone or in association with oxaliplatin, and/or irinotecan, plus either bevacizumab or cetuximab/panitumumab.

Exclusion Criteria:

* Any other malignant condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 patients with metastatic colorectal cancer treated with any fluoropyrimidine.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2019-01-16 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of C677T and A1298C MTHFR polymorphisms and overall survival | From the start date of treatment until the date of death from any cause, assessed up to 24 months
  Overall survival
Assessment of C677T and A1298C MTHFR polymorphisms and progression-free survival | From the start date of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Progression-Free survival
Assessment of C677T and A1298C MTHFR polymorphisms and response rate | From the start date of treatment until the first radiological or clinical assessment, up to 6 months.
  Response rate

SECONDARY OUTCOMES:
Assessment of C677T and A1298 MTHFR polymorphisms and toxicity | From treatment initiation to detected toxicity during treatment with any fluoropyrimidine alone or in combination with oxaliplatin, irinotecan or any biological treatment as first line therapy of colorectal metastatic cancer (up to 24 months)
  Prospective assessment of toxicity according to the National Cancer Institute Common Toxicity Criteria (NCI-CTC) 4.0 criteria according to the C677T and A1298C polymorphisms

CONTACTS AND LOCATIONS:
Overall Officials: Allan Ramos-Esquivel, Mic, Principal Investigator — Universidad de Costa Rica
Locations (1):
- Hospital San Juan de Dios, San José, Costa Rica

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramos-Esquivel A, Chinchilla-Monge R, Abbas J, Valle M. C677T and A1298C MTHFR gene polymorphisms and response to fluoropyrimidine-based chemotherapy in Mestizo patients with metastatic colorectal cancer. Pharmacogenet Genomics. 2021 Dec 1;31(9):191-199. doi: 10.1097/FPC.0000000000000440. PMID 34116533